CLINICAL TRIAL: NCT03517735
Title: Postoperative Sedation After Cardiac Surgery : Comparison Between Manual Administration and Automated Sedation
Brief Title: Automated Postoperative Sedation After Cardiac Surgery
Acronym: SEPOCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Modification of the device
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/03
Record Dates: First submitted 2018-04-19; First posted 2018-05-07 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia; Sedation; Surgery, Cardiac
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated postoperative sedation (Experimental): Automated administration of Propofol and Remifentanil.
  Interventions: Device: EasyTiva (algorithm is the property of Medsteer SAS); Drug: Propofol; Drug: Remifentanil
- Manual postoperative sedation (Active Comparator): Manual administration of Propofol and Remifentanil.
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Device: EasyTiva (algorithm is the property of Medsteer SAS) — Propofol and Remifentanil are administered automatically using a closed-loop system. Bispectral index is used as the input signal and an algorithm defines the appropriate concentrations of propofol and remifentanil. Adequate postoperative sedation is defined by a bispectral index between 55 and 75.
  Arms: Automated postoperative sedation
Drug: Propofol — The dosage is modified automatically by the device or according to the new medical prescription.
Drug: Remifentanil — The dosage is modified automatically by the device or according to the new medical prescription.

SUMMARY:
This study compares automated administration of propofol and remifentanil guided by the Bispectral index (BIS) versus manual administration for sedation after cardiac surgery.

DETAILED DESCRIPTION:
Automated sedation has the potential to improve patient care after cardiac surgery by adjusting drug doses to the minimum required for efficacy. Indeed, automated and continuous titration may avoid overdosing, improve hemodynamic stability and also decrease the mean time to tracheal extubation.

Medsteer SAS developed a controller, EasyTiva device, allowing the closed-loop coadministration of propofol and remifentanil, guided by a Bispectral Index (BIS) monitor.

Automated sedation is so facilitated by the BIS which permits continuous monitoring of electrocortical activity.

This randomized monocentric trial compares the automated administration with manual intravenous administration of propofol-remifentanil for maintaining adequate depth of hypnosis (BIS 55-75) during sedation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical procedure requiring postoperative sedation
* Low operative risk : EuroSCORE 2 ≤ 5%
* Consent for participation
* Affiliation to the social security system

Exclusion Criteria:

* Pregnant or breastfeeding women
* Neurological or muscular disorder
* Pacemaker
* Hypersensitivity to propofol or remifentanil
* Communication difficulties or neuropsychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Adequate sedation | 6 hours
  Percentage of time with BIS between 55 and 75 (BIS(55-75))

SECONDARY OUTCOMES:
Period of too deep sedation | 6 hours
  Percentage of time with BIS values less than 55
Period of too light sedation | 6 hours
  Percentage of time with BIS values greater than 75
Incidence of Burst Suppression (bsr) during sedation | 6 hours
  Presence of Burst Suppression defined by a rate > 10% for at least one minute
Level of sedation | 6 hours
  Richmond Agitation-Sedation Scale : from -5 (unarousable) to +4 (combative); the best value being 0 (alert & calm)
Level of pain during sedation | 6 hours
  Behavioral Pain Scale : from 3 (no pain) to 12 (maximum pain) 3 subscales summed :
  * Numeric Scale for Facial expression : from 1 (relaxed) to 4 (grimacing)
  * Numeric Scale for Upper limb movements : from 1 (no movement) to 4 (permanently retracted)
  * Numeric Scale for Compliance with mechanical ventilation : from 1 (tolerating movement) to 4 (unable to control ventilation)
Medical interventions | 6 hours
  Number and causes of transient or permanent interruptions in automated administration
Hemodynamic status during the sedation period | 6 hours
  Evolution of hemodynamic parameters (composite : arterial blood pressure in mmHg and heart rate in bpm)
Sedation time | 6 hours
  Duration of sedation
Delay before awakening | 6 hours
  Delay between the cessation of infusion of propofol and remifentanil and extubation.
Dose of hypnotic drug | 6 hours
  Total amount of propofol during sedation period
Dose of analgesic drug | 6 hours
  Total amount of remifentanil during sedation period
Level of consciousness after extubation | 9 hours
  Richmond Agitation-Sedation Scale : from -5 (unarousable) to +4 (combative); the best value being 0 (alert & calm)
Level of pain after extubation | 9 hours
  Behavioral Pain Scale : from 3 (no pain) to 12 (maximum pain) 3 subscales summed :
  * Numeric Scale for Facial expression : from 1 (relaxed) to 4 (grimacing)
  * Numeric Scale for Upper limb movements : from 1 (no movement) to 4 (permanently retracted)
  * Numeric Scale for Compliance with mechanical ventilation : from 1 (tolerating movement) to 4 (unable to control ventilation)
Awareness during the sedation period | 48 hours
  Awareness standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Chazot, MD, Study Chair — Hôpital FOCH
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Result] Le Guen M, Liu N, Bourgeois E, Chazot T, Sessler DI, Rouby JJ, Fischler M. Automated sedation outperforms manual administration of propofol and remifentanil in critically ill patients with deep sedation: a randomized phase II trial. Intensive Care Med. 2013 Mar;39(3):454-62. doi: 10.1007/s00134-012-2762-2. Epub 2012 Dec 6. PMID 23223772